CLINICAL TRIAL: NCT00557102
Title: Frontline Chemotherapy "Reinforced" for Cancers of the Colon and Rectum With Potentially Resectable Hepatic and/or Pulmonary Metastases: Association of FOLFIRI and ERBITUX
Brief Title: Cetuximab and Combination Chemotherapy as First-Line Therapy in Treating Patients With Colorectal Cancer That Has Spread to the Liver and/or Lung
Acronym: ERBIFORT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, France (Other Government)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000574153; CHUG-ERBIFORT; INCA-RECF0316; EUDRACT-2007-000357-54
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: liver metastases; lung metastases; recurrent rectal cancer; stage IV rectal cancer; adenocarcinoma of the rectum; adenocarcinoma of the colon; recurrent colon cancer; stage IV colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Rectal Neoplasms; Colonic Neoplasms | interventions — Cetuximab; Filgrastim; Fluorouracil; Irinotecan; Leucovorin

ARMS (1):
- cetuximab, FOLFIRI (Other)
  Interventions: Biological: cetuximab; Biological: filgrastim; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: cetuximab
Biological: filgrastim
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as irinotecan, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cetuximab together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with combination chemotherapy works as first-line therapy in treating patients with colorectal cancer that has spread to the liver and/or lung.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the tumor response rate in patients with colorectal cancer and hepatic and/or pulmonary metastases treated with cetuximab and FOLFIRI chemotherapy comprising irinotecan hydrochloride, leucovorin calcium, and fluorouracil as first-line therapy.

Secondary

* Determine the rate of resectability in patients treated with this regimen.
* Determine the overall and disease-free survival of patients treated with this regimen.
* Determine the tolerability of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive cetuximab IV over 60-120 minutes on days 1 and 8. Patients also receive FOLFIRI chemotherapy comprising irinotecan hydrochloride IV over 90 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 48 hours on days 1 and 2. Patients with 7/6 or 7/7 genotypes also receive filgrastim (G-CSF) as primary prophylaxis (patients with 6/6 genotypes receive G-CSF as secondary prophylaxis). Treatment repeats every 2 weeks for up to 8 courses in the absence of disease progression or unacceptable toxicity. Within 6 weeks after the completion of cetuximab and FOLFIRI chemotherapy, patients with responding disease undergo surgical resection of visceral metastases.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the colon or rectum
* Must have synchronous or metasynchronous unresectable hepatic metastases

  * Less than 8 hepatic metastases
  * Less than 6 segments of liver involvement with metastases
* No more than 2 potentially resectable extrahepatic (e.g., pulmonary) metastases
* Patients with visceral metastases that are potentially resectable after chemotherapy (i.e., tumor regression) are eligible
* At least 1 measurable metastasis by CT scan or MRI
* No brain metastases, bone metastases, or carcinomatous meningitis
* No celiac lymph node involvement or peritoneal cancer

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* PT rate > 70%
* Bilirubin < 30 μmol/L
* Creatinine < 130 μmol/L
* Creatinine clearance > 60 mL/min
* Not pregnant or nursing
* No other prior malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No severe unstable angina
* No symptomatic heart failure
* No other concurrent illness

PRIOR CONCURRENT THERAPY:

* At least 3 months since prior adjuvant anticancer chemotherapy
* No concurrent participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | From baseline to end of treatment

SECONDARY OUTCOMES:
Rate of resectability | From baseline to end of treatment
Overall and disease-free survival | From baseline to end of treatment
Tolerability | From baseline to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jean Marc Phelip, MD, PhD, Study Chair — University Hospital, Grenoble
Locations (1):
- CHU de Grenoble - Hopital Michallon, Grenoble, France